CLINICAL TRIAL: NCT00045708
Title: A Phase I/II Trial of BMS-247550 for Treatment of Patients With Recurrent High-grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03016; NABTT 2111; CDR257118; U01CA062475 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Giant Cell Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — ixabepilone; Anticonvulsants; Cytochrome P-450 CYP3A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A [Anticonvulsants] (Experimental): Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Pharmacological Study Phase 1
  Interventions: Drug: ixabepilone; Other: pharmacological study; Drug: Anticonvulsant
- Group B [No Anticonvulsants] (Experimental): Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Pharmacological Study Phase 1
  Interventions: Drug: ixabepilone; Other: pharmacological study
- Group C [MTD-Phase 2) (Experimental): Maximum tolerated Dose (MTD-Phase 2) - subjects treated at dose determined by Group B
  Drug: ixabepilone
  Other Names:
  BMS-247550 epothilone B lactam Ixempra Given IV
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
  Arms: Group A [Anticonvulsants]; Group B [No Anticonvulsants]
Drug: Anticonvulsant — Drugs that induce hepatic Metabolic enzymes
  Other Names: P450
  Arms: Group A [Anticonvulsants]

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. This phase I/II trial is studying the side effects and best dose of ixabepilone and how well it works in treating patients with recurrent glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of BMS-247550 when administered to adults with recurrent malignant gliomas, receiving (Group A) or not receiving (Group B) anticonvulsants known to be metabolized by the P450 hepatic enzyme complex.

II. To describe the pharmacokinetics of this route of administration, measuring BMS-247550, and determine the effects of hepatic enzyme inducing drugs, such as anticonvulsants, on the pharmacokinetics.

III. To determine the response rate of adult patients with recurrent glioma to BMS-247550 administered at the MTD.

IV. To describe the toxicity associated with this regimen in adult patients with recurrent malignant gliomas.

SECONDARY OBJECTIVES:

I. To determine the percent of patients with 6 month progression free survival, duration of progression free survival and survival associated with this therapy in adult patients with recurrent malignant gliomas.

OUTLINE: This is a phase I, dose-escalation, multicenter study followed by a phase II, safety and efficacy, multicenter study. For phase I only, patients are stratified according to cytochrome P450-inducing anticonvulsant use (yes vs no).

Phase I: Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.

Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A minimum of 10-15 patients will be accrued for the phase I portion of this study. A total of 22-33 patients will be accrued for the phase II portion of this study within 4-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven malignant glioma (anaplastic astrocytoma or glioblastoma multiforme) which is progressive or recurrent following radiation therapy +/- chemotherapy; patients with previous low grade glioma who progressed after radiotherapy +/- chemotherapy and are biopsied and found to have a high grade glioma are eligible
* Patients must have measurable progressive or recurrent malignant glioma by MRI or CT imaging
* Patients must have recovered from severe toxicity of prior therapy; an interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* HgB > 9 g/dl
* Creatinine =< 1.5mg/dl
* Total Bilirubin =< 1.5mg/dl
* Transaminases =< 2.5 times above the upper limits of the institutional norm)
* Patients must be able to provide written informed consent
* Patients must have =< 2 prior chemotherapy regimens
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; the anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant; female patients of child-bearing potential must have a negative pregnancy test
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast; patients with prior malignancies must be disease-free for >= five years
* Patients must be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment
* Patients must have a Mini Mental State Exam score of >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients with more than 2 prior chemotherapy regimens
* Patients receiving concurrent investigational agents
* Patients receiving any of the following medications which are known to be moderate to significant inhibitors of CYP3A4 are not eligible:

  * Antibiotics: clarithromycin, erythromycin, troleandomycin
  * Anti-HIV agents: delavirdine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, lopinavir
  * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200mg/day), voriconazole
  * Antidepressants: nefazodone, fluvoxamine
  * Calcium channel blockers: verapamil, diltiazem
  * Miscellaneous: amiodarone NOTE: The above list of agents was provided by the National Cancer Institute as moderate to significant inhibitors of CYP3A4 that should not be administered with BMS; there may be other agents that have similar activities on CYP3A4, however these are currently unspecified; if investigators are concerned about a particular medication's inhibitory effect on CYP3A4, they are encouraged to consult local pharmacy services for more information and to contact the principal investigator to discuss the situation further

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-seven subjects were enrolled in the Phase 1 and Phase 2 between October 2002 and November 2005. Subjects were enrolled from outpatient medical clinics
Pre-assignment Details: Please note that 4 subjects in Arm B (non-P450- 6.8mg/m2) were used in the analysis and total n for the Phase 2. Hence, 19 new subjects were accrued to the Phase 2 portion of the study at the 6.8mg/m2 dose level, but the 4 subjects already treated at 6.8gmg/m2 were included in Phase 2 analysis.
Groups:
- Group A [Anticonvulsants]; Group B [No Anticonvulsants]: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.
  Pharmacological Study
  ixabepilone: Given IV
  pharmacological study: Correlative studies
- Group 3 - MTD Phase 2: Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.
Period: Phase 1
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants] | Group 3 - MTD Phase 2
Started | 21 | 17 | 0
Completed | 21 | 16 | 0
Not Completed | 0 | 1 | 0
Not completed — early progressive disease | 0 | 1 | 0
Period: Phase 2
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants] | Group 3 - MTD Phase 2
Started | 0 | 0 | 19
Completed | 0 | 0 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A [Anticonvulsants] - Phase 1; Group B [No Anticonvulsants] - Phase 1: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.
  Pharmacological Study
  ixabepilone: Given IV pharmacological study: Correlative studies
- Phase 2: Phase II: Once the MTD is determined, additional patients receive ixabepilone at the MTD.
- Total: Total of all reporting groups
Arm/Group | Group A [Anticonvulsants] - Phase 1 | Group B [No Anticonvulsants] - Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 21 | 17 | 19 | 57
Age, Continuous [Median (Full Range); unit: years] | 53 [23 to 65] | 56 [22 to 75] | 53 [32 to 73] | 54 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 9 | 26
  Male | 16 | 5 | 10 | 31
Karnofsky Performance Status (KPS) [Number; unit: participants] — Performance status is a range where the higher score is the better score:
  100 - Normal; no complaints; no evidence of disease; 90 - Able to carry on normal activity; minor signs or symptoms of disease, 80 - Normal activity with effort; some signs or symptoms of disease; 70 - Cares for self; unable to carry on normal activity or to do active work; 60 - Requires occasional assistance, but is able to care for most of his personal needs
  participants
    60% | 2 | 3 | 0 | 5
    70% | 2 | 3 | 2 | 9
    80% | 6 | 3 | 5 | 14
    90% | 10 | 8 | 6 | 26
    100% | 1 | 0 | 6 | 7
Histology [Number; unit: participants] — pathology at time of study entry
  participants
    Glioblastoma multiforme | 15 | 14 | 14 | 46
    Malignant glioma | 1 | 0 | 1 | 2
    Anaplastic astrocytoma | 5 | 3 | 4 | 13
Anticonvulsant Use [Number; unit: participants] — subjects were either on an anticonvulsant (EIAED) enzyme inducing antiepileptic drug or on an anticonvulsant that was not enzyme inducing (-EIAED) or on NO anticonvulsant
  participants
    +EIAED | 21 | 0 | 0 | 21
    -EIAED | 0 | 12 | 10 | 25
    None | 0 | 5 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicity to Determine Maximum Tolerated Dose (MTD) of BMS-247550 in Patients With Recurrent or Progressive Malignant Glioma
Description: Starting dose for both Group A and Group B was 5mg/m2/day. A continuing reassessment method (CRM) was employed independently for each group to estimate the maximum tolerated dose. Only toxicity observed during 1st cycle of treatment (21 days) was used for dose finding. Dose limiting toxicity (DLT) defined as: ANC<500/ul, platelets<25,000, febrile neutropenia or treatment-related grade 3 or 4 non-hematologic toxicity with the exception of nausea and vomiting.
Time Frame: 21 days (1 cycle)
Population: 4 subjects from Group B (Phase 1) were included in Group 3 (Phase 2). Only those on non-anticonvulsants at the dose of 6.8mg/m2/day were treated in Phase 2. No subjects treated at the MTD for P450, as the accrual goal for phase 2 reached before MTD for p450 was determined. P450 MTD determined as 9.6mg/m2 per CRM after all enrollment of phase 2
Measure: Number; unit: DLTs
Groups:
- Group A [Anticonvulsants]; Group B [No Anticonvulsants]: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Pharmacological Study
  ixabepilone: Given IV
  pharmacological study: Correlative studies
- Group 3 - MTD (6.8mg/m2/Day) Phase 2: Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.
  ixabepilone: Given IV
  MTD for no anticonvulsant arm = 6.8mg/m2/day MTD for anticonvulsant arm = 9.6mg/m2/day
  Only no anticonvulsant subjects at 6.8mg/m2/day treated in Phase 2
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants] | Group 3 - MTD (6.8mg/m2/Day) Phase 2
Number analyzed (Participants) | 21 | 17 | 19
DLTs
  Dose level 5.0mg/m2/day | 0 | 0 | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 6.0mg/m2/day | 0 | 0 | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 6.6mg/m2/day | NA — this cohort was not tested in the anticonvulsant arm of study | 0 | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 6.8mg/m2/day | NA — this cohort was not tested in the anticonvulsant arm of study | 1 | 0
  Dose level 7.0mg/m2/day | 0 | 2 | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 7.5mg/m2/day | NA — this cohort was not tested in the anticonvulsant arm of study | 1 | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 7.7mg/m2/day | 0 | NA — this cohort was not tested in the no anticonvulsant arm of study | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 8.7mg/m2/day | 0 | NA — this cohort was not tested in the no anticonvulsant arm of study | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose Level 9.5mg/m2/day | 0 | NA — this cohort was not tested in the no anticonvulsant arm of study | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day
  Dose level 9.6mg/m2/day | 1 | NA — this cohort was not tested in the no anticonvulsant arm of study | NA — In phase 2 all subjects were treated at MTD from phase 1 group b - 6.8mg/m2/day

2. Primary Outcome: Group A (P450) Estimated MTD and Group B (nonP450) Estimated MTD of BMS-247550 in Patients With Recurrent or Progressive Malignant Glioma
Description: as for outcome 1
Time Frame: 21 days (1 cycle)
Measure: Number; unit: mg/m2/day
Groups:
- Group A [Anticonvulsants]; Group B [No Anticonvulsants]: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Pharmacological Study Phase 1
  ixabepilone: Given IV
  pharmacological study: Correlative studies
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants]
Number analyzed (Participants) | 21 | 17
mg/m2/day | 9.6 | 6.8

3. Primary Outcome: Measure Pharmacokinetic Parameters Using Estimation of Half-lives Related to BMS-247550 and Anticonvulsants
Description: T1/2,z = terminal half-life (T1/2) --- for a 2 or 3 compartment drug, idea of how long drugs stick around
Time Frame: Course 1, Day 1 (pre-infusion, midpoint of infusion, 5min prior to end of infusion, 15min, 30min, 1hr, 2hr, 3hr, 4hr and 6hr post infusion
Population: 13 of the 21 samples for P450 collected day 1 sample set and 16 of the 17 samples for the nonP40 collected day 1 sample set
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants]
Number analyzed (Participants) | 13 | 16
h | 13 (11) | 12 (3.7)

4. Primary Outcome: Measure Pharmacokinetic Parameters Using Clearance as Related to BMS-247550 and Anticonvulsant Measurements
Description: CL = clearance (how much volume of blood is cleared of the drug per unIT of time
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: l/h/m2
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants]
Number analyzed (Participants) | 13 | 16
l/h/m2 | 36 (11) | 24 (9.2)

5. Primary Outcome: Measure Pharmacokinetic Parameters Using Volume of Distribution at Steady State as Related to BMS-247550 and Anticonvulsants
Description: Vss = volume of distribution at steady-state (how widely distributed in the body the drug gets)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: l/m2
Arm/Group | Group A [Anticonvulsants] | Group B [No Anticonvulsants]
Number analyzed (Participants) | 13 | 16
l/m2 | 440 (410) | 290 (160)

6. Primary Outcome: Response Rate of Patients at the MTD
Description: Complete Response: Complete disappearance of all tumor on MRI scan, off all glucocorticoids with stable/improving neurologic exam for min4 wks.
  Partial Response: Greater than or equal to 50% reduction in tumor size on volumetric MRI scan, on a stable/decreasing dose of glucocorticoids, with stable/improving neurologic examination for min 4 wks.
  Progressive Disease: Progressive neurologic abnormalities not explained by causes unrelated to tumor progression (e.g. anticonvulsant or corticosteroid toxicity, electrolyte abnormalities, hyperglycemia, etc.) or a greater than 25% increase in the volume of the tumor by MRI scan. If neurologic status deteriorates, on stable/increasing dose of steroids, or if new lesions appear on serial MRI, further study treatment will be discontinued.
  Stable Disease: A patient whose clinical status and MRI volumetrics do not meet the criteria for Complete Response, Partial Response or Progressive Disease.
Time Frame: 3 years
Population: no objective responses observed. 19 patients treated at the MTD from during Phase 2 and 4 patients treated at the MTD during the Phase 1 nonP450 arm 2 were included in the response analysis.
Measure: Number; unit: participants
Arm/Group | Phase 2
Number analyzed (Participants) | 23
participants | 0

7. Primary Outcome: Grade 3 and 4 Toxicity (NCI Common Terminology Criteria for Adverse Events Associated With BMS-247550 Treatment in at Least 5% of Patients
Description: Proportion of patients with serious or life threatening toxicities in at least 5% of patients
Time Frame: Up to 30 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A [Anticonvulsants] - Phase 1 | Group B [No Anticonvulsants] - Phase 1 | Phase 2
Number analyzed (Participants) | 21 | 17 | 19
Participants
  Neutropenia (ANC) | 3 | 4 | 4
  WBC (leukopenia) | 1 | 3 | 4
  Hypophosphatemia (PO4) | 1 | 1 | 2
  Transfusion:pRBCs | 0 | 1 | 3
  Anemia (HGB) | 0 | 0 | 2
  Hyponatremia | 0 | 0 | 1

8. Secondary Outcome: Duration of Overall Survival
Time Frame: 1.5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A [Anticonvulsants] Phase 1: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Pharmacological Study Phase 1
- Group B [No Anticonvulsants] Phase 1: Phase I: Dose Escalation - Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 patients experience dose-limiting toxicity.
  Phase II: Once the MTD is determined, additional patients receive ixabepilone as above at the MTD.
  Pharmacological Study
  ixabepilone: Given IV
  pharmacological study: Correlative studies
Arm/Group | Group A [Anticonvulsants] Phase 1 | Group B [No Anticonvulsants] Phase 1 | Phase 2
Number analyzed (Participants) | 21 | 17 | 19
months | 4.9 [3.4 to 9.6] | 7.1 [2.9 to 15.4] | 5.8 [5.0 to 8.6]

9. Secondary Outcome: The Duration of Progression Free Survival (Phase 2)
Description: only patients treated on the nonP450 MTD
Time Frame: 1.5 years
Population: 19 patients treated at the MTD from during Phase 2 and 4 patients treated at the MTD during the Phase 1 nonP450 arm 2 were included in the response analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2: Phase II: Once the MTD is determined, additional patients receive ixabepilone at the MTD (6.8mg/m2).
Arm/Group | Phase 2
Number analyzed (Participants) | 23
months | 1.5 [1.3 to 2.3]

10. Secondary Outcome: Percent of Subjects With 6M Progression Free Survival at the Phase 2 Arm of Study
Description: subjects who are progression free at 6 month scan
Time Frame: 6 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Phase 2
Number analyzed (Participants) | 23
percent of patients | 4 [0 to 22]

ADVERSE EVENTS:
Time Frame: adverse events were collected while patients were on study and for 30 days post last day of treatment. For most patients this was 6 months. Subjects were evaluated for dose limiting toxicities (DLTs) for Phase 1 only during the first cycle (first 28 days - or until they started Cycle 2, if cycle 1 was delayed for any reason).
Arm/Group | Group A [Anticonvulsants] - Phase 1 | Group B [No Anticonvulsants] - Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/21 | 4/17 | 1/19
Other Adverse Events (participants affected / at risk) | 21/21 | 17/17 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A [Anticonvulsants] - Phase 1 (N=21) | Group B [No Anticonvulsants] - Phase 1 (N=17) | Phase 2 (N=19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decrease (Investigations) | 1 (4) | 1 (1) | 1 (1)
White blood cell decrease (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A [Anticonvulsants] - Phase 1 (N=21) | Group B [No Anticonvulsants] - Phase 1 (N=17) | Phase 2 (N=19)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (6) | 6 (6)
Anemia (HGB) (Blood and lymphatic system disorders) | 1 (1) | 11 (68) | 10 (58)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) — heartburn
Edema limbs (General disorders) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) — abdominal pain/cramping
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — (not due to neuropathy)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) — neuropathic pain
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — pneumonia
abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 4 (6) | 4 (4) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (3) | 5 (7) | 4 (5)
diarrhea (Gastrointestinal disorders) | 5 (5) | 4 (8) | 3 (3)
fatigue (General disorders) | 10 (14) | 10 (14) | 10 (13)
hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (16)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 4 (14) | 2 (7)
mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 5 (9) | 6 (7) | 7 (12)
neuropathy - sensory (Nervous system disorders) | 4 (4) | 3 (3) | 5 (6)
neutrophil count decrease (Investigations) | 5 (15) | 7 (23) | 7 (22)
platelet count decrease (Investigations) | 3 (3) | 8 (44) | 7 (30)
platelet count decrease (Investigations) | 0 (0) | 1 (13) | 1 (7)
seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (6) | 0 (0) | 2 (5)
weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
white blood cell decrease (Investigations) | 8 (26) | 10 (55) | 9 (51)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (5) | 2 (5) | 0 (0)
Aspartate aminotransferase (Investigations) | 1 (1) | 3 (4) | 1 (1)
Alanine aminotransferase (Investigations) | 0 (0) | 3 (7) | 3 (5)
hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 3 (5)

LIMITATIONS AND CAVEATS:
Phase 2 was completed using only nonP450 MTD (6.8mg/m21) as the MTD for P450 was not determined until the Phase 2 accrual had completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less